CLINICAL TRIAL: NCT04313439
Title: Targeting Taboo Thoughts In Obsessive-Compulsive Disorder Using Internet- Delivered Cognitive Therapy
Brief Title: Targeting Taboo Thoughts In Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN Dnr 2019-06047
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessions; Cognitive therapy; Internet
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Obsessive Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Online Cognitive Therapy (I-CT)
  Interventions: Other: Online cognitive therapy (I-CT)

INTERVENTIONS:
Other: Online cognitive therapy (I-CT) — The treatment is an online cognitive therapy consisting of a structured self-help program over ten weeks, divided into eight modules, administered in an encrypted web platform. The program is based on the treatment manual "The treatment of Obsessions" by Stanley Rachman. In this treatment, the participant is recommended to perform daily exercises in order to identify and modify interpretations made about the importance of their obsessive thoughts. A designated therapist have email contact with the participant within the encrypted platform.

SUMMARY:
The purpose of this pilot study is to investigate if a cognitive treatment targeting obsessive beliefs in patients with aggressive obsessions is feasible and effective as an online treatment.

DETAILED DESCRIPTION:
Patients with obsessive-compulsive disorder who presents with aggressive obsessions (also known as taboo thoughts e.g. fear of being a pedophile) and mental rituals have shown to respond less well to treatment. Thus, there is room for further innovation. The primary objective of this pilot study is to investigate if an internet-based cognitive therapy (I-CT) is feasible and effective in reducing the frequency and distress of aggressive obsessions. The study will also investigate if I-CT is associated with any significant side effects. Another objective of this study is to get a power estimate of the treatment effects for a subsequent randomized controlled study (RCT). This will be done by using an open pilot study with repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD taboo thoughts as specified in the DSM-5
* ≥ 18 years
* Situated in Sweden
* Informed consent

Exclusion Criteria:

* No signed consent
* Not fluent speaking in Swedish or cognitive abilities to read written material in the study
* Adjusted pharmacological treatment the last month symptoms that may affect OCD symptoms
* Substance dependence during the last six months
* Psychosis
* Ongoing mania or hypomania
* Suicidal risk that may affect study participation
* Personality disorder that may significantly affect the treatment participation
* Other ongoing psychological treatments that may affect OCD-symptoms
* Other primary psychiatric diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
The clinician rated Yale Brown Obsessive Compulsive Scale (Y-BOCS) | Week 0, week 10, and 6 months follow up
  Change in obsessions and compulsions from baseline to week 10 and 6 months after treatment has ended. Minimum value is 0. Maximum value is 40. Higher score means more symptoms.

SECONDARY OUTCOMES:
The self-rated Yale Brown Obsessive Compulsive Scale (Y-BOCS) | Weeks 0 to 10 through treatment and 6 months follow-up
  Change in obsessions and compulsions from baseline, during treatment to week 10 and at 6 after treatment has ended. Minimum value is 0. Maximum value is 40. Higher score means more symptoms.
Personal Significance Scale (PSS) | Weeks 0 to 10 through treatment and 6 months follow-up
  Change in perceived personal significance of intrusive thougths from baseline, during treatment to week 10 and at 6 months after treatment has ended. Minimum value is 0. Maximum value is 80. Higher score means more symptoms.
Montgomery Åsberg Depression Rating Scale - Self report (MADRS-S) | Week 0, week 10 and 6 months follow-up
  Change in depression from baseline to week 10 and at 6 months after treatment has ended. Minimum value is 0. Maximum value is 40. Higher score means more symptoms.
Clinical Global Impression (CGI) | Week 0, week 10 and 6 months follow-up
  Change in symptom severity from baseline to week 10 and 6 months after treatment has ended, and treatment response and the efficacy of treatments at week 10 and 6 months after treatment after treatment has ended. Rated by the psychologist. Minimum value is 0. Maximum value is 6. Higher score means less improvement.
Work and social adjustment scale (WSAS) | Week 0, week 10 and 6 months follow-up
  Change in functional impairment from baseline to week 10 and 6 months after treatment has ended. Minimum value is 0. Maximum value is 40. Higher score means more symptoms.
Thought Action Fusion Scale (TAFS) | Week 0, week 10 and 6 months follow-up
  Change in maladaptive cognitive intrusions from baseline to week 10 and 6 months after treatment has ended. Minimum value is 0. Maximum value is 76. Higher score means more symptoms.
Penn State Worry Questionnaire (PSWQ) | Week 0, week 10 and 6 months follow-up
  Change in worry from baseline to week 10 and 6 months after treatment has ended. Minimum value is 0. Maximum value is 80. Higher score means more symptoms.
Meta-Cognitive Questionnaire (Negative metacognitions subscale; MCQ-NC) | Week 0, week 10 and 6 months follow-up
  Change in negative meta-cognitions about worrying from baseline to week 10 and 6 months after treatment has ended. Minimum value is 0. Maximum value is 24. Higher score means more symptoms.
Patient Satisfaction Questionnaire (PSQ) | Week 10
  Satisfaction of treatment at week 10. Qualitative questions.
Adverse events (AE) | Weeks 0 to 10 through treatment and 6 months follow-up
  Number of adverse events every week during treatment and post treatment week 10.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden